CLINICAL TRIAL: NCT02542267
Title: Post-Approval Study of the GORE® VIABAHN® Endoprosthesis for the Treatment of In-Stent Restenosis (ISR) in the Superficial Femoral Artery (SFA)
Brief Title: In-Stent Restenosis Post-Approval Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISR 14-04
Record Dates: First submitted 2015-08-19; First posted 2015-09-04 (Estimated); Results first posted 2020-08-21 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Peripheral Artery Disease; Vascular Disease
Keywords: Bare Metal Stent; In-Stent Restenosis
MeSH Terms: conditions — Peripheral Arterial Disease; Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gore VIABAHN Endoprosthesis (Other): Gore VIABAHN Endoprosthesis deployed to treat failed non-covered stent(s) in the Superficial Femoral Artery
  Interventions: Device: Gore VIABAHN Endoprosthesis

INTERVENTIONS:
Device: Gore VIABAHN Endoprosthesis

SUMMARY:
The objective of the ISR 14-04 study is to evaluate post-market safety and effectiveness of GORE® VIABAHN® Endoprosthesis for treatment of In-Stent Restenosis of the Superficial Femoral Artery.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a previously implanted (> 30 days) non-covered stent(s) located in the SFA
* Patient has life-style limiting claudication, resting leg pain or minor tissue loss (Rutherford Category 2 - 5)
* Patient demonstrates an Ankle Brachial Index (ABI) <=0.9. If ABI >0.9 or not measurable, patient is eligible for study if Toe Brachial Index is <=0.5
* Patient has >=50% in-stent restenosis and / or an occlusion in a previously implanted (>30 days) non-covered stent(s) located in the superficial femoral artery defined as beginning at least 1cm below the origin of the profunda femoris artery and ending at least 1cm above the intercondylar notch.
* Patient has a maximum total lesion length of 270mm, consisting of in-stent and adjacent occlusive disease
* Patient has a reference vessel diameter between 4.0 and 6.5mm
* Patient has at least one patent infrapopliteal runoff vessel (<50% stenosis) not requiring reintervention
* Note: Additional Inclusion Criteria may apply

Exclusion Criteria:

* Patient has a known allergy to stent graft components (nickel-titanium or expanded-polytetrafluoroethylene)
* Patient has a known intolerance to anticoagulation or antiplatelet therapy
* Patient has known coagulation disorder, including hypercoagulability.
* Patient has major distal amputation (above the transmetatarsal)
* Patient has any previous surgery in the target vessel
* Patient has had previous target vessel in-stent restenosis treated by relining with another stent
* Patient has untreated flow-limiting aortoiliac stenotic disease
* Note: Additional Exclusion Criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2015-09; Primary Completion 2019-07 (Actual); Study Completion 2021-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Soukas, MD, Principal Investigator — Miriam Hospital, Providence, RI
Locations (23):
- United States (20):
  - Mount Sinai Medical Center, Miami, Florida
  - Kaiser Foundation Hospital, Honolulu, Hawaii
  - Rockford CardioVascular Associates, Rockford, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Covenant Medical Center, Inc., Saginaw, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Midwest Aortic and Vascular Institute (MAVI), North Kansas City, Missouri
  - New York University Langone Medical Center, New York, New York
  - New York Presbyterian Hospital/Weill Cornell Medical Center, New York, New York
  - North Carolina Heart and Vascular, Raleigh, North Carolina
  - Sanford Health, Fargo, North Dakota
  - Providence Heart Clinic, Portland, Oregon
  - St. Vincent's Consultants in Cardiovascular Disease, Erie, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - Greenville Hospital System, Greenville, South Carolina
  - Texas Health Research - Presbyterian Heart and Vascular, Dallas, Texas
  - Texas Health Research - Presbyterian Hospital of Plano, Plano, Texas
  - Swedish Medical Center - Heart and Vascular Research, Seattle, Washington
  - Charleston Area Medical Center, Charleston, West Virginia
- Klinikum Rosenheim, Rosenheim, Germany
- Azienda Ospedaliera Santa Maria Nuova di Reggio Emilia, Reggio Emilia, Italy
- Skånes Universitetssjukhus, Malmo, Sweden

RESULTS

PARTICIPANT FLOW:
Groups:
- Gore VIABAHN Endoprosthesis: Gore VIABAHN Endoprosthesis deployed to treat failed non-covered stent(s) in the Superficial Femoral Artery
  Gore VIABAHN Endoprosthesis
Period: Overall Study
Arm/Group | Gore VIABAHN Endoprosthesis
Started | 108
Completed | 53
Not Completed | 55
Not completed — Withdrawal by Subject | 10
Not completed — Physician Decision | 6
Not completed — Lost to Follow-up | 4
Not completed — Death | 13
Not completed — Surgical Bypass of All Study Devices | 13
Not completed — Other | 9

BASELINE CHARACTERISTICS:
Arm/Group | Gore VIABAHN Endoprosthesis
Number analyzed (Participants) | 108
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.7 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 58
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race only collected among U.S. study subjects.
  Participants
    number analyzed (Participants) | 86
    American Indian or Alaska Native | 0
    Asian | 5
    Native Hawaiian or Other Pacific Islander | 2
    Black or African American | 11
    White | 67
    More than one race | 1
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 86
  Germany | 19
  Italy | 2
  Sweden | 1
Rutherford Category [Count of Participants; unit: Participants] — Lower limb ischemia classification with 7 categories ranging from least severe (category 0) to most severe (category 6):
  Category 0 - No claudication; Category 1 - Mild claudication; Category 2 - Moderate claudication; Category 3 - Severe claudication; Category 4 - Ischemic rest pain; Category 5 - Minor tissue loss, non-healing ulcer, focal gangrene with diffuse pedal ischemia; Category 6 - Major tissue loss, extending above transmetatarsal level, functional foot no longer salvageable
  Participants
    Category 0 | 0
    Category 1 | 0
    Category 2 | 10
    Category 3 | 84
    Category 4 | 3
    Category 5 | 11
    Category 6 | 0
Ankle Brachial Index (ABI) [Mean (Standard Deviation); unit: Ratio] — The Ankle Brachial Index (ABI) is the ankle systolic pressure in the study limb divided by the highest systolic pressure in either arm. ABI values range from 0 to >1, with smaller values indicating more severe obstruction and larger values indicating better blood flow. Population: Data missing or unknown/not measured.
  Ratio
    number analyzed (Participants) | 92
    (all) | 0.670 (0.177)

OUTCOME MEASURES:

1. Primary Outcome: Primary Effectiveness
Description: Primary Effectiveness is Primary Patency defined as patent blood flow through the study device, which requires either a Peak Systolic Velocity Ratio measurement ≤ 2.5 or patent flow indicated by the Core Lab, and without repeat intervention measured at 12 months and assessed by Kaplan-Meier analysis.
Time Frame: 12 Months
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Gore VIABAHN Endoprosthesis
Number analyzed (Participants) | 108
Probability | 0.715 [0.607 to 0.797]

2. Primary Outcome: Number of Subjects Free From Procedure and Device-Related Serious Adverse Events Within 30 Days of Index Procedure
Description: Primary Safety is defined as freedom from procedure and device-related serious adverse events within 30 days of index procedure
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Gore VIABAHN Endoprosthesis
Number analyzed (Participants) | 108
Participants | 105

3. Secondary Outcome: Number of Subjects With Acute Procedural Success
Description: Acute Procedural Success is defined as successful delivery of the study device and complete coverage of the target lesion without a procedure or device-related Serious Adverse Event prior to hospital discharge.
Time Frame: During hospitalization, approximately 1-2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Gore VIABAHN Endoprosthesis
Number analyzed (Participants) | 108
Participants | 107

4. Secondary Outcome: Primary Patency at 30 Days and 12, 24, and 36 Months
Description: Primary patency is defined as patent blood flow through the study device, which requires either a PSVR measurement ≤ 2.5 or patent flow indicated by the Core Lab, without repeat intervention.
Time Frame: 30 days and 12, 24, and 36 months
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Gore VIABAHN Endoprosthesis
Number analyzed (Participants) | 108
Probability
  30 Day | 0.99 [0.932 to 0.999]
  12 Month | 0.715 [0.607 to 0.797]
  24 Month | 0.561 [0.448 to 0.661]
  36 Month | 0.449 [0.333 to 0.558]

5. Secondary Outcome: Primary Assisted Patency at 30 Days and 12, 24, and 36 Months
Description: Primary assisted patency is defined as blood flow through the study device regardless of repeat interventions to maintain patency prior to occlusion.
Time Frame: 30 days and 12, 24, and 36 months
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Gore VIABAHN Endoprosthesis
Number analyzed (Participants) | 108
Probability
  30 Day | 1.00 [1.00 to 1.00]
  12 Month | 0.772 [0.669 to 0.846]
  24 Month | 0.643 [0.529 to 0.736]
  36 Month | 0.556 [0.434 to 0.662]

6. Secondary Outcome: Secondary Patency at 30 Days and 12, 24, and 36 Months
Description: Secondary patency is defined as blood flow through the study device regardless of repeat interventions to restore patency after occlusion.
Time Frame: 30 days and 12, 24, and 36 months
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Gore VIABAHN Endoprosthesis
Number analyzed (Participants) | 108
Probability
  30 Day | 1.00 [1.00 to 1.00]
  12 Month | 0.929 [0.849 to 0.967]
  24 Month | 0.822 [0.718 to 0.891]
  36 Month | 0.732 [0.608 to 0.822]

7. Secondary Outcome: Freedom From Target Lesion Revascularization at 30 Days and 12, 24, and 36 Months
Description: Target Lesion Revascularization is defined as a repeat intervention within the study device and 5 mm proximal or distal to the edge of the study device to maintain or re-establish patency.
Time Frame: 30 days and 12, 24, and 36 months
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Gore VIABAHN Endoprosthesis
Number analyzed (Participants) | 108
Probability
  30 Day | 1.00 [1.00 to 1.00]
  12 Month | 0.828 [0.738 to 0.890]
  24 Month | 0.746 [0.645 to 0.823]
  36 Month | 0.668 [0.558 to 0.756]

8. Secondary Outcome: Freedom From Major Amputation at 30 Days and 12, 24, and 36 Months
Description: Major Amputation is defined as removal of the study limb above the metatarsals, resulting from a vascular event.
Time Frame: 30 days and 12, 24, and 36 months
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Gore VIABAHN Endoprosthesis
Number analyzed (Participants) | 108
Probability
  30 Day | 1.00 [1.00 to 1.00]
  12 Month | 1.00 [1.00 to 1.00]
  24 Month | 1.00 [1.00 to 1.00]
  36 Month | 1.00 [1.00 to 1.00]

9. Secondary Outcome: Change in Ankle Brachial Index at 30 Days
Description: The Ankle Brachial Index (ABI) is the ankle systolic pressure in the study limb divided by the highest systolic pressure in either arm. ABI values <= 0.90 are considered abnormal, 0.91-0.99 borderline, 1.00-1.40 normal, and >1.40 noncompressible. The change in ABI was measured relative to that obtained pre-procedure.
Time Frame: Pre-procedure and 30 Days
Population: Includes all subjects with Ankle Brachial Index values measured at both pre-procedure and 30 days.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Gore VIABAHN Endoprosthesis
Number analyzed (Participants) | 82
ratio
  Pre-procedure | 0.679 (0.176)
  30 Days | 1.004 (0.133)
  Change at 30 Days | 0.325 (0.205)

10. Secondary Outcome: Change in Ankle Brachial Index at 1 Year
Description: as for outcome 9
Time Frame: Pre-procedure and 1 Year
Population: Includes all subjects with Ankle Brachial Index values measured at both pre-procedure and 1 year.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Gore VIABAHN Endoprosthesis
Number analyzed (Participants) | 66
ratio
  Pre-procedure | 0.693 (0.164)
  1 Year | 0.921 (0.188)
  Change at 1 Year | 0.229 (0.235)

11. Secondary Outcome: Change in Ankle Brachial Index at 2 Years
Description: as for outcome 9
Time Frame: Pre-procedure and 2 Years
Population: Includes all subjects with Ankle Brachial Index values measured at both pre-procedure and 2 Years.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Gore VIABAHN Endoprosthesis
Number analyzed (Participants) | 54
ratio
  Pre-procedure | 0.700 (0.159)
  2 Years | 0.913 (0.187)
  Change at 2 Years | 0.213 (0.227)

12. Secondary Outcome: Change in Ankle Brachial Index at 3 Years
Description: as for outcome 9
Time Frame: Pre-procedure and 3 Years
Population: Includes all subjects with Ankle Brachial Index values measured at both pre-procedure and 3 Years.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Gore VIABAHN Endoprosthesis
Number analyzed (Participants) | 47
ratio
  Pre-procedure | 0.708 (0.162)
  3 Years | 0.937 (0.174)
  Change at 3 Years | 0.229 (0.231)

13. Secondary Outcome: Change in Rutherford Category at 30 Days
Description: The Rutherford Category is a lower limb ischemia classification with 7 categories ranging from least severe (category 0) to most severe (category 6): Category 0 - No claudication; Category 1 - Mild claudication; Category 2 - Moderate claudication; Category 3 - Severe claudication; Category 4 - Ischemic rest pain; Category 5 - Minor tissue loss, non-healing ulcer, focal gangrene with diffuse pedal ischemia; Category 6 - Major tissue loss, extending above transmetatarsal level, functional foot no longer salvageable. The change is Rutherford Category was measured relative to that obtained pre-procedure and a negative change corresponds to improved outcome.
Time Frame: Pre-procedure and 30 Days
Population: Includes all subjects with Rutherford Category measured at both pre-procedure and 30 days.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gore VIABAHN Endoprosthesis
Number analyzed (Participants) | 101
units on a scale
  Pre-procedure | 3.2 (0.7)
  30 Days | 0.6 (1.2)
  Change at 30 Days | -2.5 (1.2)

14. Secondary Outcome: Change in Rutherford Category at 1 Year
Description: as for outcome 13
Time Frame: Pre-procedure and 1 Year
Population: Includes all subjects with Rutherford Category measured at both pre-procedure and 1 year.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gore VIABAHN Endoprosthesis
Number analyzed (Participants) | 77
units on a scale
  Pre-procedure | 3.0 (0.6)
  1 Year | 0.8 (1.1)
  Change at 1 Year | -2.2 (1.3)

15. Secondary Outcome: Change in Rutherford Category at 2 Years
Description: as for outcome 13
Time Frame: Pre-procedure and 2 Years
Population: Includes all subjects with Rutherford Category measured at both pre-procedure and 2 years.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gore VIABAHN Endoprosthesis
Number analyzed (Participants) | 59
units on a scale
  Pre-procedure | 3.1 (0.6)
  1 Year | 0.6 (1.1)
  Change at 2 Years | -2.4 (1.2)

16. Secondary Outcome: Change in Rutherford Category at 3 Years
Description: as for outcome 13
Time Frame: Pre-procedure and 3 Years
Population: Includes all subjects with Rutherford Category measured at both pre-procedure and 3 years.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gore VIABAHN Endoprosthesis
Number analyzed (Participants) | 52
units on a scale
  Pre-procedure | 3.0 (0.6)
  1 Year | 0.8 (1.2)
  Change at 3 Years | -2.3 (1.5)

17. Secondary Outcome: Stent Fracture at 12, 24, and 36 Months
Description: Device stent fractures that are clearly distinguishable from previously implanted stents will be assessed by the study core lab through x-ray images.
Time Frame: 12, 24, and 36 months
Population: Includes all subjects who had x-ray or angiographic data to determine device stent fracture at the reported corresponding follow-up time period..
Measure: Count of Participants; unit: Participants
Arm/Group | Gore VIABAHN Endoprosthesis
Number analyzed (Participants) | 108
Participants
  12 Month: number analyzed (Participants) | 65
  12 Month | 0
  24 Month: number analyzed (Participants) | 54
  24 Month | 0
  36 Month: number analyzed (Participants) | 39
  36 Month | 0

ADVERSE EVENTS:
Time Frame: 36 months
Arm/Group | Gore VIABAHN Endoprosthesis
All-Cause Mortality (participants affected / at risk) | 13/108
Serious Adverse Events (participants affected / at risk) | 70/108
Other Adverse Events (participants affected / at risk) | 30/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gore VIABAHN Endoprosthesis (N=108)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Atrial fibrillation with rapid ventricular response (Cardiac disorders) | 2 (4)
Atrial flutter (Cardiac disorders) | 1 (2)
Atrioventricular junctional escape rhythm (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 2 (2)
Cardiac arrest (Cardiac disorders) | 2 (2)
Chest pain - cardiac (Cardiac disorders) | 1 (2)
Congestive cardiac failure aggravated (Cardiac disorders) | 3 (3)
Congestive heart failure (Cardiac disorders) | 2 (2)
Decompensation cardiac (Cardiac disorders) | 1 (1)
Non ST segment elevation myocardial infarction (Cardiac disorders) | 4 (5)
Non STEMI (Cardiac disorders) | 3 (3)
Paroxysmal atrial fibrillation (Cardiac disorders) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 1 (1)
Triple vessel disease (Cardiac disorders) | 1 (1)
Unstable angina (Cardiac disorders) | 2 (2)
Colon stenosis (Gastrointestinal disorders) | 1 (1)
Esophageal ulcer (Gastrointestinal disorders) | 1 (1)
Gastrointestinal bleed (Gastrointestinal disorders) | 1 (1)
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 1 (1)
Retroperitoneal bleed (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Delayed healing of wound (General disorders) | 1 (1)
In-stent arterial restenosis (General disorders) | 6 (6)
In-stent arterial stenosis (General disorders) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 2 (2)
Unknown cause of death (General disorders) | 1 (1)
Vessel puncture site hematoma (General disorders) | 2 (2)
Weakness (General disorders) | 2 (2)
Wound healing delayed (General disorders) | 1 (1)
Acute cholecystitis (Hepatobiliary disorders) | 1 (1)
Bile duct stricture (Hepatobiliary disorders) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1)
Bilateral pneumonia (Infections and infestations) | 1 (1)
Cellulitis genital organ (male) (Infections and infestations) | 1 (1)
Cellulitis of leg (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Febrile infection (Infections and infestations) | 1 (1)
Gangrene peripheral (Infections and infestations) | 1 (1)
Infectious diarrhea (Infections and infestations) | 1 (1)
Influenza A virus infection (Infections and infestations) | 1 (1)
Influenza B virus infection (Infections and infestations) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1)
Osteomyelitis of the foot (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 5 (7)
Sepsis (Infections and infestations) | 5 (8)
Urinary tract infection (Infections and infestations) | 2 (2)
Broken bones (Injury, poisoning and procedural complications) | 1 (1)
Drug overdose accidental (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2)
Fractured hip (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1)
Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 (1)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant neoplasm of hypopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Urothelial carcinoma urethra (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carotid artery disease (Nervous system disorders) | 1 (1)
Cerebral hemorrhage (Nervous system disorders) | 1 (1)
Cerebral infarct (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (2)
Grand mal seizure (Nervous system disorders) | 1 (1)
Hemiparesis (left) (Nervous system disorders) | 1 (1)
Internal carotid artery stenosis (Nervous system disorders) | 1 (1)
Ischemic stroke (Nervous system disorders) | 1 (1)
Near syncope (Nervous system disorders) | 1 (1)
Seizures (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 3 (3)
Subarachnoid hemorrhage (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 1 (1)
Tremor aggravated (Nervous system disorders) | 1 (1)
Device occlusion (Product Issues) | 18 (22)
Thrombosis in device (Product Issues) | 5 (6)
Mental status changes (Psychiatric disorders) | 1 (2)
Acute kidney failure (Renal and urinary disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Acute retention of urine (Renal and urinary disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 1 (1)
Vaginal prolapse (Reproductive system and breast disorders) | 1 (1)
Acute on chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive airways disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary necrotizing granuloma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Foot ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Acute limb ischemia (Vascular disorders) | 2 (2)
Aortic stenosis (Vascular disorders) | 1 (1)
Atherosclerosis (Vascular disorders) | 1 (1)
Critical limb ischemia (Vascular disorders) | 1 (4)
Hypertensive crisis (Vascular disorders) | 1 (1)
Hypertensive emergency (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (3)
Malignant hypertension (Vascular disorders) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gore VIABAHN Endoprosthesis (N=108)
In-stent arterial restenosis (General disorders) | 14 (20)
Device occlusion (Product Issues) | 12 (12)
Arterial stenosis (Vascular disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and Investigator agree not to submit any Publication until Study Completion and the multi-center Publication has been published. If the multi-center Publication has not been submitted within 12 months of Study Completion, Institution and Investigator may be able to proceed with submission of the Publication.

DOCUMENTS (2):
  • Study Protocol (2015-12-10): https://cdn.clinicaltrials.gov/large-docs/67/NCT02542267/Prot_000.pdf
  • Statistical Analysis Plan (2015-05-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT02542267/SAP_001.pdf